CLINICAL TRIAL: NCT00650819
Title: A Multicenter, Double-blind, Randomized, Active-controlled Parallel Groups Study Comparing The Efficacy and Safety of The Daily Co-Administration of Ezetimibe 10 mg With Simvastatin 20 mg Vs Simvastatin Or Ezetimibe Alone in Subjects With Primary Hypercholesterolemia
Brief Title: Comparison of Ezetimibe Plus Simvastatin Versus Ezetimibe or Simvastatin Alone in Subjects With Primary Hypercholesterolemia (Study P03757)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P03757
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe, Simvastatin Drug Combination; Ezetimibe; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ezetimibe + Simvastatin (Experimental)
  Interventions: Drug: Ezetimibe + Simvastatin
- Simvastatin (Active Comparator)
  Interventions: Drug: Simvastatin
- Ezetimibe (Active Comparator)
  Interventions: Drug: Ezetimibe

INTERVENTIONS:
Drug: Ezetimibe + Simvastatin — ezetimibe 10 mg plus simvastatin 20 mg once daily for 8 weeks
  Other Names: SCH 58235
  Arms: Ezetimibe + Simvastatin
Drug: Simvastatin — simvastatin 20 mg plus ezetimibe placebo once daily for 8 weeks
  Arms: Simvastatin
Drug: Ezetimibe — Ezetimibe 10 mg plus simvastatin placebo once daily for 8 weeks
  Other Names: SCH 58235
  Arms: Ezetimibe

SUMMARY:
This is a multicenter, randomized, double blind; active-controlled parallel groups study enrolling subjects with primary hypercholesterolemia. Subjects receive ezetimibe, simvastatin, or the combination once daily for 8 weeks to determine the effect on LDL-cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Subjects must be >= 18 years and <= 75 years of age.
* Subjects with Primary Hypercholesterolemia must be finished the Lab test listed below and the results must be available at the time of randomization at Visit 3 (Baseline Visit).

  * LDL-C concentration > 3.64 mmol/L (140mg/dL) to <= 6.3 mmol/L (250 mg/dL) using the Friedewald calculation
  * Total cholesterol (TC) > 5.2mmol/L (200mg/dL) to < 12.7mmol/L (500mg/dL)
  * Triglyceride concentrations of <= 3.99 mmol/L (350 mg/dL)
  * Liver transaminases (ALT, AST) must be within normal limits, with no active liver disease and CK < 50% above the upper limit of normal
  * Clinical laboratory tests (CBC, blood chemistries, urinalysis) must be within normal limits
* Subjects must report a stable weight history for at least 4 weeks prior to entry into study at Visit 3 (Baseline Visit).
* Women of childbearing potential (includes women who are less than 1 year postmenopausal and women who become sexually active) must be using an acceptable method of birth control (e.g. medically prescribed IUD, condom in combination with spermicide) or be surgically sterilized (e.g., hysterectomy or tubal ligation).
* Subjects must be free of any clinically significant diseases other than hyperlipidemia that would interfere with study evaluations.
* Subjects must understand and be able to adhere to the dosing and visit schedules, and must agree to remain on a cholesterol-lowering diet for the duration of the study.

Exclusion Criteria:

* Subjects whose body mass index (BMI = weight [kg]/height2 [m]) is >= 30 Kg/m^2 at Visit 3 (Baseline Visit).
* Subjects who have known hypersensitivity to HMG-CoA reductase inhibitors.
* Subjects who consume > 14 alcoholic drinks per week. (A drink is: a can of beer, glass of wine, or single measure of spirits).
* Any condition or situation, which in the opinion of the investigator, might pose a risk to the subject or interfere with participation in the study.
* Women who are pregnant or nursing
* Subjects who have not observed the designated washout periods for any of the prohibited medications outlined in protocol
* Congestive heart failure defined by NYHA as Class III or IV.
* Uncontrolled cardiac arrhythmia.
* Myocardial infarction, coronary bypass surgery or angioplasty within 6 months of study entry.
* Unstable or severe peripheral artery disease within 3 months of study entry.
* Unstable angina pectoris within 6 months of study entry.
* Uncontrolled hypertension (treated or untreated) with systolic blood pressure > 160 mm Hg or diastolic > 100 mm Hg of study entry.
* Uncontrolled (as determined by HbA1c > 7 %) or newly diagnosed (within 1month of study entry) diabetes mellitus.
* Uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins, i.e., secondary causes of hyperlipidemia, such as secondary hypercholesterolemia due to hypothyroidism (TSH above upper limit of normal). Subjects with a history of hypothyroidism who are on a stable therapy of thyroid hormone replacement for at least 6 weeks are eligible for enrollment if TSH levels are within normal limits before enrollment.
* Known Impaired renal function (plasma creatinine > 2.0 mg/dL), or nephrotic syndrome of study entry.
* Disorders of the hematologic, digestive, or central nervous systems including cerebrovascular disease and degenerative disease that would limit study evaluation or participation.
* Known HIV positive.
* Cancer within the past 5 years (except for successfully treated basal and squamous cell carcinomas).
* History of mental instability, drug/alcohol abuse within the past 5 years, or major psychiatric illness not adequately controlled and stable on pharmacotherapy.
* Subjects with known coagulopathy (PT and PTT at Visit 1 >1.25 times control)
* Women receiving hormonal therapy, including hormone replacement, any estrogen antagonist/agonist, or oral contraceptives.
* Any other condition which in the opinion of the investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in and completing the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2004-06-01 (Actual); Primary Completion 2005-02-01 (Actual); Study Completion 2005-02-01 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in LDL-C concentration. | 8 weeks

SECONDARY OUTCOMES:
Percent change from baseline in total cholesterol, triglycerides, and HDL-C. | 8 weeks